CLINICAL TRIAL: NCT05083936
Title: Prospective Comparison of 18F-FDG and 18F-FET PET for Response Evaluation in Patients With Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Minyoung Oh, Assistant professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FET-PCNSL
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Patients With Suspected or Diagnosed Central Nervous System Lymphoma
MeSH Terms: interventions — (18F)fluoroethyltyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]FET PET (Experimental)
  Interventions: Drug: [18F]FET

INTERVENTIONS:
Drug: [18F]FET — Imaging evaluation using LAT1/4F2hc substrate overexpressed in brain tumor
  Other Names: Fluoroethyl-L-tyrosine

SUMMARY:
The overall goal of this imaging trial is to prospectively compare the usefulness of 18F-FDG PET and 18F-FET PET in evaluating treatment response and predicting prognosis in patients with central nervous system lymphoma.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

* Be ≥ 19 years of age.
* Patients diagnosed with central nervous system lymphoma by surgery/biopsy or suspected of central nervous system lymphoma by anatomical imaging examination such as MRI.
* Patients who have results or are planning to examine 18F-FDG PET in the above patients.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject fulfil any single criteria described below:

* Pediatric and adolescent patients under 19 years of age.
* The patient is pregnant, is attempting to become pregnant, or is nursing (breast-feeding) to children.
* Patients with diagnosed or suspected lymphoma lesions in organs other than the cetral nervous system.
* Based on the investigator's judgement, if the patient makes it impossible to collect complete data for a clinical trial due to personal or other reasons.
* Patients who cannot stably have PET/CT due to claustrophobia, dyskinesia, anxiety disorder, seizure, etc.
* Based on the investigator's judgement, if the patient has a serious and/or uncontrolled and/or unstable medical disease (e.g., congestive heart failure, acute myocardial infarction, severe lung disease, chronic renal disease or chronic liver disease, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of target to background ratio between baseline, mid-therapy and end-of treatment PET in patients with primary central nervous system lymphoma | 20-40 minutes post injection

SECONDARY OUTCOMES:
1.5 year progression free survival | 18months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu, South Korea